CLINICAL TRIAL: NCT02517177
Title: Alterations in Autonomic Cardiovascular Control Induced at Partial G Forces
Acronym: AUTOCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-008
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular parameters measurements (Other)
  Interventions: Other: Parabolic flight; Other: Cardiovascular parameters measurements

INTERVENTIONS:
Other: Parabolic flight
Other: Cardiovascular parameters measurements

SUMMARY:
As a direct consequence of exposure to microgravity, astronauts experience a number of physiological changes which can lead to serious medical implications. Most immediate and significant is the headward shift of body fluids and the removal of gravitational loading from bone and muscles, resulting in progressive changes of the cardiovascular and musculoskeletal systems. The cardiovascular systems is subject to rapid changes which has been demonstrated in studies of short term (shuttle) and long term missions to Skylab and MIR.

Our main hypothesis is that there is a linear relationship between the gravity level (0G, 0.16G, 0.38G, 1G, 1.8G) and the cardiovascular parameters (heart rate (HR), heart rate variability (HRV), blood pressure and blood pressure variability (BPV) as well the spectral analysis of HRV and BPV.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteer
* aged from 20 to 35
* affiliated to a Social Security system and, for non-French resident, holding an European Health Insurance Card (EHIC)
* who accepts to take part in the study
* who has given their written stated consent
* who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude .There will be no additional test

Exclusion Criteria:

* persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated,
* persons who take any medication or drugs influencing the autonomic cardiovascular control

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The heart rate (HR) and the heart rate variability (HRV) derived from the ECG | baseline
The systolic, diastolic and mean arterial blood pressure (SP, DP, MAP) | baseline
The autonomic cardiovascular control evaluated with a spectral analysis of HRV and BPV. | baseline
the blood pressure variability (BPV) derived from the continuous blood pressure recording | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France